CLINICAL TRIAL: NCT04966559
Title: Effects of a Peripherally Acting µ-opioid Receptor Antagonist on Recurrent Acute Pancreatitis An Investigator-initiated, Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Effects of a Peripherally Acting µ-opioid Receptor Antagonist on Recurrent Acute Pancreatitis
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Collaborators: Odense University Hospital (Other); Hvidovre University Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Chief Physician, MD, PhD, DMSc, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAMORA_RAP; 2021-000069-34 (EudraCT Number); N-20210034 (Other: North Denmark Region Committee in Health Research Ethics)
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis | interventions — naldemedine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo treatment (Placebo Comparator): Film-coated matched placebo-tablets consisting of:
  Core:
  Mannitol, USP/Ph. Eur./JP Croscarmellose Sodium, NF/Ph. Eur./JP Magnesium Stearate, NF/Ph. Eur./JP
  Coating:
  Opadry Yellow Purified Water, USP/EP
  Interventions: Drug: Placebo treatment
- Naldemedine treatment (Active Comparator): Film-coated matched active-tablets consisting of:
  Core:
  Naldemedine Tosylate (0,2 mg) Mannitol, USP/Ph. Eur./JP Croscarmellose Sodium, NF/Ph. Eur./JP Magnesium Stearate, NF/Ph. Eur./JP
  Coating:
  Opadry Yellow Purified Water, USP/EP
  Interventions: Drug: Naldemedine 0.2 MG Oral Tablet

INTERVENTIONS:
Drug: Placebo treatment — Active drug/placebo is handed out equivalent of 1 tablet of 0,2 mg Naldemedine or placebo daily for 365 days.
  Arms: Placebo treatment
Drug: Naldemedine 0.2 MG Oral Tablet — Active drug/placebo is handed out equivalent of 1 tablet of 0,2 mg Naldemedine or placebo daily for 365 days.
  Arms: Naldemedine treatment

SUMMARY:
This study will investigate the effect of a peripheral acting opioid antagonist (PAMORA) on the disease course of patients with recurrent acute inflammation of the pancreas (acute pancreatitis). The study will be conducted by treating outpatients suffering from recurrent acute pancreatitis with a PAMORA (naldemedine) for 12 months.

DETAILED DESCRIPTION:
In this study, the effects of a peripheral acting µ-opioid receptor antagonist (PAMORA) on disease recurrence and progression in patients with recurrent acute pancreatitis (RAP) will be investigated. Patients with RAP will be administered 0,2 mg naldemedine orally daily or matching placebo. This medication is defined as the investigational product. Naldemedine is approved by the European Medical Agency for treatment of opioid-induced constipation. This PAMORA have not previously been investigated in patients with pancreatitis. The dose regimes for this study will be according to label. It has previously been shown, in patients with opioid-induced obstipation and healthy subjects, that opioid antagonism incl. PAMORA treatment increases gut motility, relaxes gastrointestinal sphincters, increases the intestinal water content and improves the immune response, without affecting analgesia. The affinity of PAMORAs to the µ-opioid receptors is much stronger than opioid analgesics. Therefore, they as antagonists have the potential to counteract the harmful effects of opioids on the gut mucosa, bacterial translocation and inflammation despite the high levels of exogenous opioids present in patients with pancreatitis. PAMORAs do not cross the blood-brain barrier and consequently do not interfere with analgesia or other central effects of opioids.

It is hypothesized that treatment with the PAMORA naldemedine will antagonize the harmful effects of opioids without reducing analgesia in patients with RAP and hence reduce disease severity and improve clinical outcomes. If successful, this study will for the first time document the effects of a targeted pharmacotherapy in RAP with the potential benefit of improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study specific procedures
* Able to read and understand Danish or Swedish (depending on site)
* Male or female age between 18 and 74 years
* At least one attack of non-biliary AP (as defined by the revised Atlanta criteria) within the last 12 months and at least two attacks within 5 years
* Clinically stable at time of inclusion
* The researcher believes that the participant understands what the study entails, is capable of following instructions, can attend when needed, and is expected to complete the study
* The investigator will ensure that fertile female participants have a negative pregnancy test before treatment initiation and use contraception during the study period. The following methods of contraception, if properly used, are generally considered reliable: oral contraceptives, patch contraceptives, injection contraceptives, vaginal contraceptive ring, intrauterine device, surgical sterilization (bilateral tubal ligation), vasectomized partner, double barrier (condom and pessary), or sexual abstinence. Methods of contraception will be documented in the source documents

Exclusion Criteria:

* Known allergy towards study medication
* Known or suspected major stenosis or perforation of the intestines
* Known or suspected abdominal cancer (incl. intestine, pancreas and the biliary tree)
* Pre-existing renal insufficiency (defined as habitual eGFR below 45)
* Female participants that are lactating
* Severe pre-existing comorbidities (assessed by investigator upon inclusion)
* Attack of AP requiring admission within two weeks prior to inclusion
* Gallstone etiology of RAP (MRCP or endoscopic ultrasound excluding biliary etiology of AP must be available prior to enrolment as part of the protocol)
* Treatment with potent CYP3A4-inhibitors (ketoconazol, itraconzol, ritonavir) or P-gp inhibitors (e.g. cyclosporine).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of AP attacks verified by the Atlanta Criteria | Observation period starts from day of randomization and ends after a minimum of 6 months and a maximum of 12 months
  The primary outcome is defined as time to (recurrent) AP attack(s) verified by the Atlanta Criteria between the naldemedine group and the placebo group.
  The Atlanta Criteria is the current gold standard for the diagnosis of AP attack, and it requires a minimum of two out three of the following features:
  (i) Abdominal pain typical for acute pancreatitis featuring acute onset of a severe and persistent epigastric pain radiating to the back (ii) Serum amylase levels > three times greater than the normal upper limit (iii) Findings of pancreatic inflammation in contrast-enhanced computed tomography, magnetic resonance imaging or transabdominal ultrasonography.

SECONDARY OUTCOMES:
Pain intensity | Observation period starts from day of randomization and ends after a minimum of 6 months and a maximum of 12 months
  Individual difference between subgroups in number and severity of pain attacks (without fulfilling AP criteria) assessed by pain diary and modified Brief Pain Inventory short form on visual analogue scale from 0-10 (0 is no pain and 10 is worst pain). For each attack, participants will be asked to fill in the pain attack diary and the modified Brief Pain Inventory short form once.
Gut function (BSFS) | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in gut function assessed by The Bristol Stool Form Scale for assessment of stool frequency as well as stool consistency (scale from 1-7, where 1 is firmeste and 7 is softest).
Gut function (GSRS) | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in gut function assessed by Gastrointestinal Symptom Rating Scale which is a disease-specific instrument of 15 items combined into five symptom clusters depicting reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Health resource utilization | Observation period starts from day of randomization and ends after a minimum of 6 months and a maximum of 12 months
  Difference in health resource utilization (measured in frequency and type of health services used (e.g. blood sample, MRI etc.) that can be converted into danish currency for economic analyses) between subgroups based on service codes (all services have unique service codes stored digitally).
Pancreatic volume | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference in pancreatic volume measured in cubic centimeters cm^3 between subgroups, measured by MRI.
Exocrine pancreatic function | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in exocrine pancreatic function assessed by fecal-elastase (µg/g) test.
Endocrine pancreatic function | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in endocrine pancreatic function assessed by hemoglobinA1c (HbA1c) (mmol/mol) test.
Quality of life (EORTC QLQ-C30) | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in quality of life assessed by EORTC QLQ-C30 questionnaire. The questionnaire has been validated for assessment of quality of life in patients with chronic pancreatitis and is composed of single-item measures and multi-item scales with scores ranging from 0 to 100 after linear transformation of the raw score. A high score for a functional scale represents a high level of functioning, as does a high score for the global health status, while a high score for the symptom items represents a high level of symptomatology.
Impression of change | Day of randomization and at follow up visit after a minimum of 6 months and a maximum of 12 months
  Difference between subgroups in Patient Global Impression of Change. PGIC is a seven-point rating scale for self-report of a patient's experienced efficacy of treatment on their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M. Drewes, Professor, Principal Investigator — Aalborg University Hospital
Locations (5):
- Denmark (4):
  - Mech-Sense, Department of Medical Gastroenterology, Aalborg University Hospital, Aalborg, Jutland
  - Digestive Disease Center K, Bispebjerg University Hospital, Bispebjerg
  - Gastrounit, Hvidovre University Hospital, Hvidovre
  - Odense Pancreas Center, Svendborg
- Karolinska University Hospital, Stockholm, Solna (l1:00), Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Cook ME, Knoph CS, Davidsen L, Frokjaer JB, Bruun NH, Novovic S, Hadi A, Jorgensen MT, Mortensen MB, Schaffalitzky O, Nielsen LBJ, Berner-Hansen M, Drewes AM, Olesen SS. Naldemedine for the Prevention of Recurrent Acute Pancreatitis: A Randomised, Double-Blind, Placebo-Controlled Trial. United European Gastroenterol J. 2026 Feb;14(1):e70178. doi: 10.1002/ueg2.70178. PMID 41553774
- [Derived] Cook ME, Knoph CS, Fjelsted CA, Frokjaer JB, Bilgrau AE, Novovic S, Jorgensen MT, Mortensen MB, Nielsen LBJ, Hadi A, Berner-Hansen M, Rutkowski W, Vujasinovic M, Lohr M, Drewes AM, Olesen SS. Effects of a peripherally acting micro-opioid receptor antagonist for the prevention of recurrent acute pancreatitis: study protocol for an investigator-initiated, randomized, placebo-controlled, double-blind clinical trial (PAMORA-RAP trial). Trials. 2023 May 1;24(1):301. doi: 10.1186/s13063-023-07287-z. PMID 37127657